CLINICAL TRIAL: NCT04686383
Title: A Phase I, Multi-center, Open-label, Dose-escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of CAL056 Mesylate in Patients With Solid Tumors Resistant or Refractory to Standard Treatments
Brief Title: Safety, Tolerability, and Pharmacokinetics of CAL056 Mesylate in Patients With Resistant or Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Calgent Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CAL056-101
Record Dates: First submitted 2020-12-15; First posted 2020-12-28 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Resistant or Refractory Solid Tumors
Keywords: CAL056 mesylate; Oncology; Dose-limiting toxicity; Maximum tolerated dose; Pharmacokinetics; Safety
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1: 20 mg CAL056 mesylate (Experimental): Patients will receive oral dose of 20 mg CAL056 mesylate once daily under fasting condition in the morning for 28 days during each cycle.
  Interventions: Drug: CAL056 mesylate
- Cohort 2: 40 mg CAL056 mesylate (Experimental): Patients will receive oral dose of 40 mg CAL056 mesylate once daily under fasting condition in the morning for 28 days during each cycle.
  Interventions: Drug: CAL056 mesylate
- Cohort 3: 80 mg CAL056 mesylate (Experimental): Patients will receive oral dose of 80 mg CAL056 mesylate once daily under fasting condition in the morning for 28 days during each cycle.
  Interventions: Drug: CAL056 mesylate
- Cohort 4: 120 mg CAL056 mesylate (Experimental): Patients will receive oral dose of 120 mg CAL056 mesylate once daily under fasting condition in the morning for 28 days during each cycle.
  Interventions: Drug: CAL056 mesylate
- Cohort 5: 160 mg CAL056 mesylate (Experimental): Patients will receive oral dose of 160 mg CAL056 mesylate once daily under fasting condition in the morning for 28 days during each cycle.
  Interventions: Drug: CAL056 mesylate

INTERVENTIONS:
Drug: CAL056 mesylate — Dosage form: 20 mg CAL056 mesylate/tablet

SUMMARY:
This is a multi-center, open-label, dose-escalation, phase I study to evaluate the safety, tolerability, pharmacokinetics (PK), preliminary efficacy, and pharmacodynamics of CAL056 mesylate in cancer patients with resistant or refractory solid tumors.

DETAILED DESCRIPTION:
Patients with resistant or refractory malignant solid tumors and no standard treatment available will be screened for the eligibility. Patients will be screened within 28 days prior to the first dose of CAL056 mesylate. Eligible patients will receive CAL056 mesylate daily with the assigned dose level for 28 days (Day 1 to Day 28) for each treatment cycle. Patients will be administered with CAL056 mesylate at clinical site at scheduled visits (i.e. Day 1/Visit 1, Day 8/Visit 2, Day 15/ Visit 3, Day 22/Visit 4, Day 28/Visit 5). Remaining doses of CAL056 mesylate on all other days will be self-administered by patients at home. After the administration of CAL056 mesylate on Day 1 and Day 28, patients can stay at the clinical site for 24 hours to have safety monitoring and blood samples collected for PK analysis.

Only patients completing Cycle 1 without a dose-limiting toxicity (DLT) or disease progression will be allowed to continue the subsequent cycles at the same dose level. The maximum number of dosing cycle is 6 cycles in each patient in this study. Continuation of using CAL056 mesylate may be permitted after the evaluation of the risk/benefit in individual patient by the Investigators and with the approval of Calgent.

During the Cycle 1 of study period, a total of 5 visits are scheduled to evaluate the safety, PK, preliminary efficacy, and pharmacodynamics of CAL056 mesylate. Each visit is planned on Day 1 of each subsequent cycle if patients continue the treatment of CAL056 mesylate. After the end treatment of CAL056 mesylate, an end of treatment (EOT) visit and a safety follow-up visit will be scheduled.

ELIGIBILITY:
Inclusion Criteria:

* Patients with age ≥ 18 years old
* Patients with resistant or refractory solid tumors confirmed by histology which are unresponsive to standard therapies
* Patients with at least one measurable lesion per RECIST version 1.1.
* Patients with Eastern Cooperative Oncology Group performance status (ECOG-PS) ≤ 2
* Patients with at least 3 months of life expectancy as judged by the investigators
* Patients with adequate bone marrow reserve and organ function
* Patients with the negative result for testing Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2)
* Female patients are eligible to participate if they are of non-childbearing potential or have documentation of a negative serum pregnancy test at screening. Sexually active pre-menopausal women of childbearing potential must agree to use adequate, highly effective contraceptive measures during and upon completion of the study and for at least 6 months after the last dose of study drug
* Male patients who agree to use an adequate method of contraception during and upon completion of the study and for at least 6 months after the last dose of study drug
* Patients must be willing and be able to provide written informed consent for the study.

Exclusion Criteria:

* History of other invasive malignancy that is currently active and/or has been treated within 12 months prior to screening
* Patients with the presence of symptomatic central nervous system (CNS) metastases requiring radiation treatment, surgery, or continuous use of corticosteroids or patients with untreated or developing brain metastasis causing any symptoms, such as neurologic deficits, seizures, or headache
* Any prior adjuvant cytotoxic chemotherapy within 4 weeks prior to screening
* Any radiotherapy within 2 weeks prior to screening
* Pre-existing chemotherapy-related peripheral neuropathy
* Currently participating or has participated in a study of an investigational product within 4 weeks prior to the first dose of CAL056 mesylate
* Patients with history of organ or stem cell transplant requiring immunosuppressive medications
* Active autoimmune disease
* Pulmonary conditions such as sarcoidosis, silicosis, idiopathic pulmonary fibrosis, or hypersensitivity pneumonitis
* Patients who have chronic obstructive pulmonary disease (COPD) or asthma
* Has a history of pneumonitis that required steroids or current pneumonitis
* Known significant liver disease
* Known history of human immunodeficiency virus (HIV) infection (HIV 1/2 antibodies)
* Has received live attenuated vaccination within 30 days prior to the first dose of CAL056 mesylate
* Female patients who is pregnant, breast-feeding, or planning to become pregnant
* Patients with corrected QT interval (QTc) interval of > 450 msec.
* Has history of clinically significant or severe gastrointestinal disease or condition that may affect drug absorption within the past 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-12-29 (Actual); Primary Completion 2022-06-07 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events (AEs), serious adverse events (SAEs), and treatment emergent adverse events (TEAEs) | From screening visit until safety follow-up visit (at 28 days after the EOT) or before starting new anticancer treatment, whichever comes first (up to 1-year)
  To evaluate the safety and tolerability of CAL056 mesylate in cancer patients.
Number of patients with AEs qualified as dose-limiting toxicities (DLTs) | Cycle 1 (28 days)
  Dose-limiting toxicities are evaluated using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Determination of tolerability and maximum tolerated dose (MTD) of CAL056 mesylate by DLTs using NCI CTCAE version 5.0 | Cycle 1 (28 days)
  MTD will be the highest dose associated with occurrence of DLTs ≤ 33% (e.g. 2/6 evaluable patients experience a DLT during the first treatment Cycle).
Evaluation of the PK profile of CAL056 mesylate: Maximum observed concentration (Cmax) | At Day 1 and Day 28 of Cycle 1, at Day 1 of subsequent cycles until Cycle 6 (except for Cycle 2) (each cycle is 28 days in length)
  Pharmacokinetics profile will be evaluated following a comprehensive PK parameter, such as Cmax.
Evaluation of the PK profile of CAL056 mesylate: Time to reach Cmax (Tmax) | At Day 1 and Day 28 of Cycle 1, at Day 1 of subsequent cycles until Cycle 6 (except for Cycle 2) (each cycle is 28 days in length)
  Pharmacokinetics profile will be evaluated following comprehensive PK parameter, such as Tmax.
Evaluation of the PK profile of CAL056 mesylate: Apparent terminal elimination half-life (t½) | At Day 1 and Day 28 of Cycle 1, at Day 1 of subsequent cycles until Cycle 6 (except for Cycle 2) (each cycle is 28 days in length)
  Pharmacokinetics profile will be evaluated following comprehensive PK parameter, such as t½.
Evaluation of the PK profile of CAL056 mesylate: Area under the concentration-time curve (AUC) | At Day 1 and Day 28 of Cycle 1, at Day 1 of subsequent cycles until Cycle 6 (except for Cycle 2) (each cycle is 28 days in length)
  Pharmacokinetics profile will be evaluated following a comprehensive PK parameter, AUC.
Preliminary determination of the recommended phase II dose (RP2D) of CAL056 mesylate | Cycle 1 (28 days)
  The RP2D will be preliminarily determined by the PK profile, type and severity of drug related toxicity, clinical suitability for long-term administration.

SECONDARY OUTCOMES:
Evaluation of the preliminary efficacy of CAL056 mesylate in tumor response as assessed by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 | At the screening visit and within 7 days prior to Day 1 of odd cycles (i.e., Cycle 3 and Cycle 5) (each cycle is 28 days in length) and at EOT/Early Termination (ET) (up to 21 months)
  Tumor response will be assessed by RECIST version 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Yun Yen, M.D., Study Chair — Calgent Biotechnology Co., Ltd
Locations (3):
- United States (2):
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - NEXT Oncology, 2829 Babcock Road Suite 300, San Antonio, Texas
- Tzu Chi General Hospital, Taipei Branch, New Taipei City, Taiwan